CLINICAL TRIAL: NCT04083638
Title: Investigation of the Relationship Between Erythrocyte Transfusion and Nutrition and Necrotizing Enterocolitis in Preterm Infants: a Randomized Controlled Clinical Trial
Brief Title: The Relationship Between Erythrocyte Transfusion and Nutrition and Necrotizing Enterocolitis in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Senem Alkan Özdemir, MD, Associate Professor of Neonatology, Dr. Behcet Uz Children's Hospital
Other Study IDs: 2019/279
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Necrotizing Enterocolitis of Newborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Control group
  Interventions: Diagnostic Test: IFAB
- Group 2: Feeding will not stop during the transfusion
  Interventions: Diagnostic Test: IFAB

INTERVENTIONS:
Diagnostic Test: IFAB — Intestinal Fatty Acid Binding Protein will be taken from all participants before the tx and after the tx

SUMMARY:
In this study; The aim of this study was to investigate the changes in fasting and dietary and mesenteric blood flow in the acute period during and after transfusion and to evaluate the necrotizing enterocolitis.

ELIGIBILITY:
Inclusion Criteria:

* <32 gestational week and/or <1500 g birth weight

Exclusion Criteria:

* Major congenital anomalies, hemodynamic instability

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants
Sampling Method: Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
necrotizing enterocolitis | 0-48 hours after tx
Mortality | 0-24 hour after tx
  If all babies die after tx study will be finished

CONTACTS AND LOCATIONS:
Overall Officials: Rüya Çolak, MD, Study Chair — Behcet Uz Children's Hospital
Locations (1):
- Behçet Uz Children's Hospital, İzmirli, İzmir, Turkey (Türkiye)